CLINICAL TRIAL: NCT04944537
Title: Current Situation and Analysis of ICU Management in Severe Trauma Patients: A Survey From 12 Provinces in China
Brief Title: Current Situation and Analysis of ICU Management for Severe Trauma Patients in China
Acronym: NJJLISTP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lulu Gu (Other)
Responsible Party: Sponsor-Investigator, Lulu Gu, specialist nurse, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Other Study IDs: 20210615; 18CXZ040 (Other Grant/Funding Number: Xianghong Ye)
Record Dates: First submitted 2021-06-15; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: ICU; Trauma Injury; ICU Acquired Weakness
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU management for patients with severe trauma: Group to investigate the current status of ICU management for patients with severe trauma
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Over the past 10 years, there has not been a consensus on ICU nursing management based on the concept of injury control. Case management for patients with serious trauma continues to be initiated in general services and after discharge.There is no critical care unit case management strategy for the high-risk population following acute intake. Consequently, there is an urgent need to develop and enhance ICU nursing best practice after injury control.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses, doctors, and rehabilitation technicians on the job;
* Formally hired, and working in ICU for more than 6 months, with ICU patient management experience;
* Voluntary participation in this survey.

Exclusion Criteria:

* retirees, interns/nurses/rehabilitation technicians, staff on leave, regular training doctors, and departmental nurses;
* those who are unwilling to participate in this survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Formally hired, and working in ICU for more than 6 months, with ICU trauma patient management experience
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-06-27 (Estimated); Study Completion 2021-12-27 (Estimated)

PRIMARY OUTCOMES:
Cognition of ICU severe trauma patient | 20 days
  The management status of severe trauma patients: including 5 dimensions of risk factor management, related complications management, ICU transition ward preparation plan, discharge preparation plan, and doctor-patient communication

CONTACTS AND LOCATIONS:
Overall Officials: Xianghong Ye, Principal Investigator — Jinling Hosp Res Inst of general surgery,Nanjing Univ,Sch Med
Locations (1):
- Jinling Hosp Res Inst of general surgery,Nanjing Univ Sch Med, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li ZL, Jin P, Yuan HH, Xu JF, Chen YJ, Wang ZQ, Li Z, Fang Y, Yu XD. Regional whole-course trauma care - Experiences from a county-level hospital. Chin J Traumatol. 2018 Oct;21(5):250-255. doi: 10.1016/j.cjtee.2018.08.001. Epub 2018 Aug 24. PMID 30270142
- [Background] Antunes PSL, LibOrio PR, Shimoda GM, Pivetta LGA, Parreira JG, Assef JC. Trauma Quality Indicators' usage limitations in severe trauma patients. Rev Col Bras Cir. 2021 Feb 24;48:e20202769. doi: 10.1590/0100-6991e-20202769. eCollection 2021. PMID 33656134
- [Background] Coccolini F, Kluger Y, Moore EE, Maier RV, Coimbra R, Ordonez C, Ivatury R, Kirkpatrick AW, Biffl W, Sartelli M, Hecker A, Ansaloni L, Leppaniemi A, Reva V, Civil I, Vega F, Chiarugi M, Chichom-Mefire A, Sakakushev B, Peitzman A, Chiara O, Abu-Zidan F, Maegele M, Miccoli M, Chirica M, Khokha V, Sugrue M, Fraga GP, Otomo Y, Baiocchi GL, Catena F; WSES Trauma Quality Indicators Expert Panel. Trauma quality indicators: internationally approved core factors for trauma management quality evaluation. World J Emerg Surg. 2021 Feb 23;16(1):6. doi: 10.1186/s13017-021-00350-7. PMID 33622373
- [Background] Tahan HM, Kurland M, Baker M. Understanding the Increasing Role and Value of the Professional Case Manager: A National Study From the Commission for Case Manager Certification: Part 1. Prof Case Manag. 2020 May/Jun;25(3):133-165. doi: 10.1097/NCM.0000000000000429. PMID 32235196
- [Background] Jeppesen E, Iversen VV, Hansen IS, Reierth E, Wisborg T. Trauma research in the Nordic countries, 1995-2018 - a systematic review. Scand J Trauma Resusc Emerg Med. 2020 Mar 12;28(1):20. doi: 10.1186/s13049-020-0703-6. PMID 32164776